CLINICAL TRIAL: NCT04043000
Title: Effects of Super 13 Pro & Prebiotics on the Human Intestinal Microflora: a Double-blind, Randomized, Placebo-controlled Study
Brief Title: Super 13 Pro & Prebiotics on the Human Intestinal Microflora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Super13-2019
Record Dates: First submitted 2019-07-10; First posted 2019-08-02 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Probiotics; Prebiotics
Keywords: Prebiotics; Probiotics; Microbiota
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: This study aim to investigate the roles of the test article in improving gastrointestinal functions and gut microbiota of humans. A total 40 healthy adults were recruited and randomly divided into experimental and control groups, with 20 subjects each, for a 4-week trial. The subjects took the test article, "Super 13 Pro & Prebiotics" or the control article, "The placebo without Super 13 Pro & Prebiotics" during the 4-week drug-intake period. Fecal specimens were collected at the 0th, 2nd, and 4th weeks of the trial for analyzing the bacterial counts of Bifidobacterium spp., Clostridium perfringens, Lactobacillus spp., and Coliform.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subjects took the test article, "Super 13 Pro & Prebiotics" or the control article, "The placebo without Super 13 Pro & Prebiotics" during the 4-week drug-intake period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Super 13 Pro & Prebiotics (Experimental): "Super 13 Pro & Prebiotics" was given three times a day for four weeks.
  Interventions: Dietary Supplement: Super 13 Pro & Prebiotics
- Placebo (Placebo Comparator): " The placebo without Super 13 Pro & Prebiotics" was given three times a day for four weeks.
  Interventions: Dietary Supplement: Super 13 Pro & Prebiotics

INTERVENTIONS:
Dietary Supplement: Super 13 Pro & Prebiotics — "Super 13 Pro & Prebiotics" was given three times a day for four weeks.

SUMMARY:
This study aim to investigate the roles of the test article in improving gastrointestinal functions and gut microbiota of humans. A total 40 healthy adults were recruited and randomly divided into experimental and control groups, with 20 subjects each, for a 4-week trial. The subjects took the test article, "Super 13 Pro & Prebiotics" or the control article, "The placebo without Super 13 Pro & Prebiotics" during the 4-week drug-intake period. Fecal specimens were collected at the 0th, 2nd, and 4th weeks of the trial for analyzing the bacterial counts of Bifidobacterium spp., Clostridium perfringens, Lactobacillus spp., and Coliform.

DETAILED DESCRIPTION:
This study aim to investigate the roles of the test article in improving gastrointestinal functions and gut microbiota of humans. A total 40 healthy adults were recruited and randomly divided into experimental and control groups, with 20 subjects each, for a 4-week trial. The subjects took the test article, "Super 13 Pro & Prebiotics" or the control article, "The placebo without Super 13 Pro & Prebiotics" three times a day during the 4-week drug-intake period. Fecal specimens were collected at the 0th, 2nd, and 4th weeks of the trial for analyzing the bacterial counts of Bifidobacterium spp., Clostridium perfringens, Lactobacillus spp., and Coliform.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers and willing to give voluntary written informed consent

Exclusion Criteria:

* Major systemic disease
* Pregnancy, parturient and feeding woman, or expect to be pregnant
* Abnormal liver function
* Abnormal renal function
* Abnormal gastrointestinal function
* Take medications for gastrointestinal and metabolic diseases
* Occurrences of severe diseases within 6 months, such as stroke, myocardial infarction, major trauma and surgery • Poor compliance for study protocol

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Intestinal Microflora: Bifidobacterium spp. | 2nd, and 4th weeks
  Change from baseline bacterial counts at 2nd, and 4th weeks. Fecal specimens were collected at the 0th, 2nd, and 4th weeks of the trial for analyzing the bacterial counts.
Intestinal Microflora: Clostridium perfringens | 2nd, and 4th weeks
  Change from baseline bacterial counts at 2nd, and 4th weeks. Fecal specimens were collected at the 0th, 2nd, and 4th weeks of the trial for analyzing the bacterial counts.
Intestinal Microflora: Lactobacillus spp. | 2nd, and 4th weeks
  Change from baseline bacterial counts at 2nd, and 4th weeks. Fecal specimens were collected at the 0th, 2nd, and 4th weeks of the trial for analyzing the bacterial counts.
Intestinal Microflora: Coliform | 2nd, and 4th weeks
  Change from baseline bacterial counts at 2nd, and 4th weeks. Fecal specimens were collected at the 0th, 2nd, and 4th weeks of the trial for analyzing the bacterial counts.

CONTACTS AND LOCATIONS:
Overall Officials: YI-HSIEN LIN, Principal Investigator — Cheng-Hsin General Hospital
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taipei City, Taiwan